CLINICAL TRIAL: NCT00074022
Title: A Phase I/2 Study of GTI-2040 Combined With Docetaxel In Metastatic Or Unresectable Locally Advanced Non-Small Cell Lung Cancer
Brief Title: GTI-2040 and Docetaxel in Treating Patients With Recurrent, Metastatic, or Unresectable Locally Advanced Non-Small Cell Lung Cancer, Prostate Cancer, or Other Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02563; PMH-PHL-017; N01CM17107 (NIH); CDR0000341677 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Recurrent Prostate Cancer; Stage III Prostate Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer; Stage IV Prostate Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms | interventions — GTI2040; Docetaxel

ARMS (1):
- Treatment (GTI-2040, docetaxel) (Experimental): Phase I (closed to accrual as of 8/5/2004): Patients receive GTI-2040 IV continuously on days 1-14. Patients also receive docetaxel IV over 1 hour on day 3 during course 1 and on day 1 for all subsequent courses. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of GTI-2040 and docetaxel until the MTD is determined. The MTD is defined as the dose at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. The RP2D is defined as the dose preceding the MTD.
  Phase II: Patients receive GTI-2040 and docetaxel at the RP2D as in phase I.
  Interventions: Biological: GTI-2040; Drug: docetaxel; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: GTI-2040 — Given IV
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase I/II trial to study the effectiveness of combining GTI-2040 with docetaxel in treating patients who have recurrent, metastatic, or unresectable locally advanced non-small cell lung cancer, prostate cancer, or other solid tumors. GTI-2040 may stop the growth of cancer cells by blocking the enzymes necessary for their growth. It may also increase the effectiveness of docetaxel by making the tumor cells more sensitive to the drug. Combining GTI-2040 with docetaxel may kill more tumor cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the recommended phase II dose of GTI-2040 and docetaxel in patients with recurrent, metastatic, or unresectable locally advanced non-small cell lung cancer, prostate cancer, or other solid tumors (phase I study closed to accrual as of 8/5/2004).

II. Determine the toxicity of this regimen in these patients. III. Determine the objective tumor response rate in patients treated with this regimen.

IV. Determine the stable disease rate, time to disease progression, objective response duration, and duration of stable disease in patients treated with this regimen.

V. Determine the pharmacokinetics of GTI-2040 when administered in combination with docetaxel in these patients.

VI. Correlate the pharmacokinetics of GTI-2040 with the biological and toxic effects of this regimen in these patients.

VII. Correlate baseline and post-treatment levels of ribonucleotide reductase activity in tumor biopsies and peripheral blood mononuclear cells and tumoral expression of c-myc, ras, pRAF1, pMAPK, and markers of apoptosis with clinical outcome in patients treated with this regimen.

OUTLINE: This is an open-label, dose-escalation, multicenter study.

Phase I (closed to accrual as of 8/5/2004): Patients receive GTI-2040 IV continuously on days 1-14. Patients also receive docetaxel IV over 1 hour on day 3 during course 1 and on day 1 for all subsequent courses. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of GTI-2040 and docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. The recommended phase II dose (RP2D) is defined as the dose preceding the MTD.

Phase II: Patients receive GTI-2040 and docetaxel at the RP2D as in phase I.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 12-48 patients (12-18 for phase I [closed to accrual as of 8/5/2004] and 15-30 for phase II) will be accrued for this study within 4-16 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of 1 of the following:

  * Solid tumor malignancy (phase I only)*
  * Prostate cancer (phase I only)*
  * Non-small cell lung cancer (phase I and II)*
* Recurrent, metastatic, locally advanced unresectable, or treatment-refractory disease
* Measurable disease

  * At least 1 unidimensionally measurable lesion at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * Previously irradiated lesions are considered measurable provided they have demonstrated progression before study entry
  * No bone-only disease

    * Must have measurable disease other than bone lesions
* No stage IIIA or IIIB non-small cell lung cancer without a malignant pleural or pericardial effusion that is eligible for first-line radical combined chemotherapy and radiotherapy
* No known progressive or symptomatic brain metastases

  * Asymptomatic brain metastases allowed
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 3 months
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No history of coagulopathy
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 2 times ULN (3.5 times ULN if liver metastases are present)
* INR no greater than 1.3
* APTT no greater than 1.25 times ULN
* Creatinine no greater than 1.5 times ULN
* Creatinine clearance at least 50 mL/min
* No symptomatic congestive heart failure
* No evidence of cardiac dysfunction
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active peptic ulcer disease
* No poorly controlled diabetes mellitus
* No pre-existing grade 2 or greater neuropathy
* No ongoing or active infection
* No contraindication to corticosteroids
* No psychiatric illness or social situation that would limit compliance with study requirements
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to study drugs
* No other concurrent uncontrolled illness
* One, and only one, prior chemotherapy regimen for advanced disease (not including adjuvant therapy) allowed

  * Neoadjuvant/adjuvant chemotherapy allowed
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin) and recovered
* Prior multiple lines of endocrine therapy for advanced solid tumors allowed
* More than 4 weeks since prior endocrine therapy and recovered
* Concurrent steroids allowed
* See Disease Characteristics
* More than 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy to sole site of measurable disease
* Prior surgery allowed
* No concurrent anticoagulant therapy

  * Concurrent low-dose warfarin for central line thrombosis prophylaxis allowed
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational or commercial agents or therapies intended to treat the malignancy
* Concurrent bisphosphonates allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2003-10; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing dose limiting toxicities (DLTs), graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) v2.0 (Phase I) | Up to day 21
Objective tumor response as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) (Phase II) | Up to day 42
  The 95% confidence intervals will be provided.

SECONDARY OUTCOMES:
Stable disease rate | Up to 6 weeks
Response duration | Up to 4 years
  The 95% confidence intervals will be provided.
Toxicities of GTI-2040 combined with docetaxel, graded according to the NCI CTC v2.0 | Up to 4 years
Time to disease progression | Up to 4 years
Duration of stable disease | Up to 6 weeks
Level of ribonucleotide reductase (RNR) activity | Up to week 10
  Logistic regression and descriptive statistics will be used.
Tumoral expression in terms of c-myc, R2 subunit protein levels and markers of proliferation (cyclin B1) and apoptosis (activated caspase 3) | Up to week 10
  Logistic regression and descriptive statistics will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Leighl, Principal Investigator — Princess Margaret Hospital Phase 2 Consortium
Locations (1):
- Princess Margaret Hospital Phase 2 Consortium, Toronto, Ontario, Canada